CLINICAL TRIAL: NCT01294007
Title: A Radiographic Analysis Using PureGen Osteoprogenitor Cell Allograft Versus Autologous Bone in Posterolateral Fusion in a Side-by-Side Comparison in the Same Patient (PLF)
Brief Title: Radiographic Analysis Using PureGen Versus Autologous Bone in Posterolateral Fusion (PLF)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Product no longer on the market
Sponsor: Alphatec Spine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-000061
Record Dates: First submitted 2011-02-09; First posted 2011-02-11 (Estimated); Results first posted 2022-10-05 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-09

CONDITIONS: Lumbar Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

ARMS (2):
- Study Graft Composite (Experimental): AlphaGraft ProFuse Demineralized Bone Scaffold are soaked in PureGen according to Preparation for Use and handling technique. The graft composite is placed on the randomized study side contralateral to the autograft bone graft per surgeon's standard technique for PLF. The wound is closed according to surgeon's standard technique.
  Post operative care will be according to the site specific standard of care. An avoidance of heavy physical activity and limitations on working, lifting, bending etc. are common precautions post procedure. The decision to use a post operative orthosis is left to the discretion of the Investigator.
  Interventions: Biological: PureGen Osteoprogenitor Cell Allograft
- Control Graft Composite (Active Comparator): Contralateral to the study graft composite, placement of posterolateral fusion graft composite containing iliac crest bone (5 cc/level/side) and local autograft composite (equal volume split with study side). Supplemental posterior pedicle screw fixation utilizing Zodiac, Illico or Xenon Spinal Fixation system.
  * A defined volume of iliac crest bone graft (indicated in table 2) is harvested and combined with 50% of the previously harvest morselized local bone
  * The graft composite is placed on the randomized control side using standard technique for PLF
  Interventions: Procedure: Autograft bone

INTERVENTIONS:
Biological: PureGen Osteoprogenitor Cell Allograft — PureGen Osteoprogenitor Cell Allograft with posterior transpedicular fixation.
  Arms: Study Graft Composite
Procedure: Autograft bone — Iliac Crest and Local Autograft Bone
  Arms: Control Graft Composite

SUMMARY:
The purpose of this study is to evaluate the rate and quality of fusion of PureGen Osteoprogenitor Cell Allograft, compared to autograft bone in instrumented posterolateral fusion (PLF) procedures.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational, self-control study assessing screened and consented subjects undergoing instrumented posterolateral fusion for degenerative disc disease (DDD) at 1 to 2 contiguous levels between L1 and S1.

Patients diagnosed with DDD will be screened for enrollment based on inclusion and exclusion criteria outlined in this protocol. Subjects who are successfully screened and sign an informed consent will undergo PLF surgery utilizing PureGen, Alphagraft ProFuse Demineralized Bone Scaffold (DBS), and ZODIAC, Illico, or Xenon Fixation system (pedicle screw and rod fixation system)

Subjects will be followed at 6 weeks, 3, 6, 12 and 24 month post-operative visits. Standard radiographs will be taken at these visits to evaluate fusion rate and quality. Oswestry Disability Index (ODI) and Visual Analog Scale (VAS) self-assessment questionnaires and neurological exams will be administered to measure pain and function scores. A computerized tomography (CT) scan will be taken at the 6-month to further assess rate and quality of fusion. A conditional 12 and 24 month post operative CT may also be taken. Procedure related and PureGen related adverse events will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lumbar degenerative disc disease in up to two contiguous levels between L1 and S1
* Subjects with back and/or leg pain indicated for posterior stabilization with or without decompression at any level and posterolateral fusion (PLF)
* Unresponsive to conservative treatment for at least 6 months
* Radiographic evidence of primary diagnosis

Exclusion Criteria:

* More than 2 levels requiring posterolateral fusion
* Spondylolisthesis greater than Grade I
* Prior failed fusion surgery at any lumbar level(s)
* Systemic or local infection in the disc or cervical spine, past or present
* Active systemic disease
* Osteoporosis, osteomalacia, or other metabolic bone disease that would significantly inhibit bone healing
* Use of other bone graft, Bone Morphogenetic Protein (BMP) or bone graft substitutes in addition to or in place of those products specified
* BMI greater than 40
* Use of post operative Spinal Cord Stimulator (SCS)
* Known or suspected history of alcohol and/or drug abuse
* Involved in pending litigation or worker's compensation related to the spine
* Pregnant or planning to become pregnant during the course of the study
* Insulin-dependent diabetes mellitus
* Life expectancy less than duration of study
* Any significant psychological disturbance that could impair consent process or ability to complete self-assessment questionnaires
* Undergoing chemotherapy or radiation treatment, or chronic use of oral or injected steroids or prolonged use of non-steroidal anti-inflammatory drugs.
* Known history of hypersensitivity or anaphylactic reaction to dimethyl sulfoxide (DMSO)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beverly Hills, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Enrollment: Single patient enrolled for site
Period: Overall Study
Arm/Group | Patient Enrollment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No controls were included.
Groups:
- Study Graft Composite: AlphaGraft ProFuse Demineralized Bone Scaffold are soaked in PureGen according to Preparation for Use and handling technique. The graft composite is placed on the randomized study side contralateral to the autograft bone graft per surgeon's standard technique for PLF. The wound is closed according to surgeon's standard technique.
  Post operative care will be according to the site specific standard of care. An avoidance of heavy physical activity and limitations on working, lifting, bending etc. are common precautions post procedure. The decision to use a post operative orthosis is left to the discretion of the Investigator.
  PureGen Osteoprogenitor Cell Allograft: PureGen Osteoprogenitor Cell Allograft with posterior transpedicular fixation.
- Control Graft Composite: Contralateral to the study graft composite, placement of posterolateral fusion graft composite containing iliac crest bone (5 cc/level/side) and local autograft composite (equal volume split with study side). Supplemental posterior pedicle screw fixation utilizing Zodiac, Illico or Xenon Spinal Fixation system.
  * A defined volume of iliac crest bone graft (indicated in table 2) is harvested and combined with 50% of the previously harvest morselized local bone
  * The graft composite is placed on the randomized control side using standard technique for PLF
  Autograft bone: Iliac Crest and Local Autograft Bone
- Total: Total of all reporting groups
Arm/Group | Study Graft Composite | Control Graft Composite | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Age, Continuous [Mean (Full Range); unit: years] | 71 |  | 71
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Fusion
Description: Number of patients with fusion at the 6- and conditional 12- and 24-month visit
Time Frame: 6, 12 and 24 month
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Enrollment
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Arm/Group | Patient Enrollment
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No